CLINICAL TRIAL: NCT05503979
Title: Eliminación de la infección Por el Virus de la Hepatitis C en PWID en Los Estados Del Norte de México
Brief Title: Elimination of Hepatitis C Virus Among Users of Substances
Acronym: EHCUS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Graciela Elia Castro Narro, Principal Investigator, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Other Study IDs: GAS-3800-21-22-1
Record Dates: First submitted 2022-08-03; First posted 2022-08-17 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Hepatitis C in Substance Users
Keywords: HCV; Elimination; Substance Users
MeSH Terms: interventions — Sofosbuvir; velpatasvir; sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A blood sample will be taken for HCV detection by PCR (polymerase chain reaction)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Substances Users: Substances users confirmed with Viral Load for HCV. after that will be evaluated through laboratory studies (CBC and blood chemistry), HIV/HBV (Hepatitis B Virus) serology, fibrosis status will be evaluated through APRI (AST to Platelet Ratio Index) and FIB-4. The antiviral treatment (sofosbuvir/Velpatasvir) will be chosen according to the characteristics of each patient and follow-up will be maintained according to the national plan with a visit at the end of treatment and 12 weeks after its end to assess SVR. The importance of this project is characterized by minimal monitoring, patients and doctors education by telementoring, multidisciplinary teams and integral treatment.
  Interventions: Drug: Sofosbuvir 400 MG / Velpatasvir 100 MG [Epclusa]

INTERVENTIONS:
Drug: Sofosbuvir 400 MG / Velpatasvir 100 MG [Epclusa] — 1 tab every 24 hrs for 12 weeks
  Other Names: Epclusa

SUMMARY:
Substance users are a vulnerable group that should be prioritized in HCV (Hepatitis C Virus) elimination efforts in Mexico and in which it is feasible to carry out micro-elimination programs. It is an important group to treat both because of its high prevalence and because of the dynamic spread of infection among the general population. HCV seropositivity has not been documented in this group of people in Mexico City, the metropolitan area and the northern states of the country, nor has the sustained viral response been evaluated in this group of patients in the Mexican population.

DETAILED DESCRIPTION:
The investigators would use a work team, the program and the value proposal would be presented to the local authorities, the coordinator of the national commission against dependencies and doctors. The investigators would use an algorithm designed for the first-step diagnosis of HCV in SUs (Substances Users) , and defined the key centers for screening and linking to care.

The project is planned as follows:

* Screening: SUs in centers of substance users in Mexico City, the metropolitan area and states in the North of the country will be evaluated with rapid tests. Those with a positive result will be selected.
* Diagnosis: Patients with a positive rapid test result will undergo a viral load test against HCV. Those with positive results will be selected.
* Link-up: Those who are confirmed positive will be profiled to receive treatment at INCMNSZ. they will receive damage reduction to prevent reinfection or primary infection in negatives (granted by the rehabilitation center).
* Treatment: The treatment will be received in a certified hospital (INCMNSZ) to treat patients with HCV infection, the treatment will be indicated by doctors who work in this hospital in the treatment consultations for hepatitis C or in centers with substance users with doctors trained to administer the treatment. This training will be received by telementoring. And also during the treatment, follow-up will be given with telementoring sessions if necessary. This group of people has personality characteristics that require a integral treatment, so it will be a integral and multidisciplinary treatment with psychological care and harm reduction (provided by the rehabilitation center)
* Confirm SVR: A viral load test will be performed 12 weeks after the end of treatment to corroborate SVR. They will be given after this a mentorship for harm reduction and advice against reinfections

The importance of this project is characterized by minimal monitoring, patients and doctors education by telementoring, multidisciplinary teams and integral treatment

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years.
* Active infection by hepatitis C virus.
* People who use substances and who are users of rehabilitation centers in Mexico City, the metropolitan area and the northern states of the country.
* Signature of informed consent

Exclusion Criteria:

* all those who do not fit the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Substances Users who are registered in the rehabilitation centers that comply with the applicable regulations in Mexico City, the metropolitan area and the northern states of the country.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-11-15 (Estimated); Primary Completion 2023-08-15 (Estimated); Study Completion 2024-05-15 (Estimated)

PRIMARY OUTCOMES:
Sustained viral response (SVR) in people who use substances in the Mexico City metropolitan area and the northern states of the country. | through study completion, an average of 1 year
  Number por participants who achive SVR whit the treatment

SECONDARY OUTCOMES:
Seroprevalence and prevalence of HCV in people who use substances in the Mexico City metropolitan area and the northern states of the country. | through study completion, an average of 1 year
  Number of participants with chronic HCV infection
No Sustained viral response (SVR) in people who use Substances in the Mexico City | through study completion, an average of 1 year
  Number of participants who does not achive RVS

CONTACTS AND LOCATIONS:
Overall Officials: Graciela Castro-Narro, MD, Principal Investigator — INCMNSZ

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication would be shared
Supporting Information: CSR
Time Frame: By 2024, once the enrollment of patients and the analyzes have been completed, this publication will be published and can be consulted
Access Criteria: An Open Access journal will be searched so that the information can be consulted

REFERENCES:
- [Background] Yehia BR, Schranz AJ, Umscheid CA, Lo Re V 3rd. The treatment cascade for chronic hepatitis C virus infection in the United States: a systematic review and meta-analysis. PLoS One. 2014 Jul 2;9(7):e101554. doi: 10.1371/journal.pone.0101554. eCollection 2014. PMID 24988388
- [Background] Mendizabal M, Alonso C, Silva MO. Overcoming barriers to hepatitis C elimination. Frontline Gastroenterol. 2019 Jul;10(3):207-209. doi: 10.1136/flgastro-2018-101114. Epub 2019 Feb 1. No abstract available. PMID 31288259
- [Background] Lazarus JV, Safreed-Harmon K, Thursz MR, Dillon JF, El-Sayed MH, Elsharkawy AM, Hatzakis A, Jadoul M, Prestileo T, Razavi H, Rockstroh JK, Wiktor SZ, Colombo M. The Micro-Elimination Approach to Eliminating Hepatitis C: Strategic and Operational Considerations. Semin Liver Dis. 2018 Aug;38(3):181-192. doi: 10.1055/s-0038-1666841. Epub 2018 Jul 9. PMID 29986353
- [Background] Wansom T, Falade-Nwulia O, Sutcliffe CG, Mehta SH, Moore RD, Thomas DL, Sulkowski MS. Barriers to Hepatitis C Virus (HCV) Treatment Initiation in Patients With Human Immunodeficiency Virus/HCV Coinfection: Lessons From the Interferon Era. Open Forum Infect Dis. 2017 Feb 11;4(1):ofx024. doi: 10.1093/ofid/ofx024. eCollection 2017 Winter. PMID 28480293
- [Background] Vandenbroucke JP, von Elm E, Altman DG, Gotzsche PC, Mulrow CD, Pocock SJ, Poole C, Schlesselman JJ, Egger M; STROBE Initiative. Strengthening the Reporting of Observational Studies in Epidemiology (STROBE): explanation and elaboration. Int J Surg. 2014 Dec;12(12):1500-24. doi: 10.1016/j.ijsu.2014.07.014. Epub 2014 Jul 18. PMID 25046751
- See also: Global Health Sector Strategy for Viral Hepatitis 2016-2021: Ending Viral Hepatitis. — https://apps.who.int/iris/handle/10665/250578